CLINICAL TRIAL: NCT02771691
Title: Efficacy of Mentalization-Based Group Therapy for Adolescents: A Pilot Randomised Controlled Trial
Brief Title: Mentalization-Based Group Therapy for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELHF10-595
Record Dates: First submitted 2016-04-25; First posted 2016-05-13 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2017-11

CONDITIONS: Deliberate Self-Harm
Keywords: Adolescent
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBT therapy plus treatment as usual (Experimental): Mentalization based group treatment for adolescents plus standard care
  Interventions: Other: Mentalization-Based Group Therapy for Adolescents
- Treatment as usual alone (No Intervention): Standard care provided by local Child and Adolescent Mental Health Services

INTERVENTIONS:
Other: Mentalization-Based Group Therapy for Adolescents
  Arms: MBT therapy plus treatment as usual

SUMMARY:
This is a prospective parallel group design of group-based Mentalization-Based Therapy for Adolescents (MBT-A) through a pilot randomised controlled trial comparing group-based MBT-A plus treatment as usual (TAU) to TAU alone. As a pilot study, we aim to determine: the effectiveness of our recruitment strategies; compliance with protocol/procedures; trends towards reduced self-harm.

ELIGIBILITY:
Inclusion Criteria:

* Self-harm behaviour in the past 6 months
* In receipt of treatment from local Child and Adolescent Mental Health Services
* Competent and willing to provide written, informed consent.

Exclusion Criteria:

* Severe learning disability or pervasive developmental disorder
* Acute psychotic episode
* Eating disorder in the absence of self-harm.
* Non-English speaking
* Current involvement in other ongoing treatment research

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Self-harm as measured by the self-harm sub scale of the Risk-taking and Self-harm Inventory for Adolescents (Vrouva et al, 2010) | 12 weeks
Self-harm and related hospital use as reported in National Health Service patient records | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CAMHS, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Griffiths H, Duffy F, Duffy L, Brown S, Hockaday H, Eliasson E, Graham J, Smith J, Thomson A, Schwannauer M. Efficacy of Mentalization-based group therapy for adolescents: the results of a pilot randomised controlled trial. BMC Psychiatry. 2019 Jun 6;19(1):167. doi: 10.1186/s12888-019-2158-8. PMID 31170947